CLINICAL TRIAL: NCT03174041
Title: A 4-Part Phase 1 Study to Evaluate the Effect of GDC-0853 on the Pharmacokinetics of Midazolam, Rosuvastatin, and Simvastatin and the Effect of Itraconazole on the Pharmacokinetics of GDC-0853
Brief Title: A Drug-Drug Interaction Study Between GDC-0853 and Midazolam, Itraconazole, Rosuvastatin, and Simvastatin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: GP39616
Record Dates: First submitted 2017-05-04; First posted 2017-06-02 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Healthy Participants
MeSH Terms: interventions — Midazolam; fenebrutinib; Rosuvastatin Calcium; Simvastatin; Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1 (Experimental): Participants will receive a single dose of midazolam followed by multiple doses of GDC-0853 coadministered with a single dose of midazolam.
  Interventions: Drug: Midazolam; Drug: GDC-0853; Drug: Midazolam and GDC-0853
- Part 2 (Experimental): Participants will receive a single dose of rosuvastatin followed by multiple doses of GDC-0853 coadministered with a single dose of rosuvastatin.
  Interventions: Drug: GDC-0853; Drug: Rosuvastatin; Drug: Rosuvastatin and GDC-0853
- Part 3 (Experimental): Participants will receive a single dose of simvastatin followed by multiple doses of GDC-0853 coadministered with a single dose of simvastatin.
  Interventions: Drug: GDC-0853; Drug: Simvastatin; Drug: Simvastatin and GDC-0853
- Part 4 (Experimental): Participants will receive a single dose of GDC-0853 followed by multiple doses of itraconazole coadministered with a single dose of GDC-0853.
  Interventions: Drug: GDC-0853; Drug: Itraconazole; Drug: GDC-0853 and itraconazole

INTERVENTIONS:
Drug: Midazolam — Single dose midazolam
  Arms: Part 1
Drug: GDC-0853 — Multiple doses GDC-0853 for 6 days
  Arms: Part 1; Part 2; Part 3
Drug: Midazolam and GDC-0853 — Multiple doses GDC-0853 and single dose midazolam
  Arms: Part 1
Drug: Rosuvastatin — Single dose rosuvastatin
  Arms: Part 2
Drug: Rosuvastatin and GDC-0853 — Multiple doses GDC-0853 and single dose rosuvastatin
  Arms: Part 2
Drug: Simvastatin — Single dose simvastatin
  Arms: Part 3
Drug: Simvastatin and GDC-0853 — Multiple doses GDC-0853 and single dose simvastatin
  Arms: Part 3
Drug: GDC-0853 — Single dose GDC-0853
  Arms: Part 4
Drug: Itraconazole — Multiple doses itraconazole for 6 days
  Arms: Part 4
Drug: GDC-0853 and itraconazole — Multiple doses itraconazole and single dose GDC-0853
  Arms: Part 4

SUMMARY:
The purpose of this study is to assess the potential for a drug interaction between GDC-0853 and midazolam, itraconazole, rosuvastatin, and simvastatin.

DETAILED DESCRIPTION:
This will be a 4-part study, with each part being an open-label fixed-sequence evaluation conducted in healthy adult participants. Approximately 64 participants will be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

* Within body mass index range of 18 to 31 kilograms per square meter, inclusive
* Females will be non-pregnant, non-lactating, and either postmenopausal or surgically sterile
* Males will either be sterile or agree to use an approved method of contraception

Exclusion Criteria:

* Significant history or clinical manifestation of any significant metabolic, allergic/immunologic/immunodeficiency, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, or psychiatric disorder (as determined by the investigator)
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the investigator
* Participation in any other investigational study drug trial in which receipt of any investigational study drug occurred within 30 days or 5 half-lives, whichever is longer, prior to check in
* History of malignancy, except for appropriately treated carcinoma in situ of the cervix or non-melanoma skin carcinoma with 3-year disease-free follow up
* Any acute or chronic condition or any other reason that, in the opinion of the investigator, would limit the participant's ability to complete and/or participate in this clinical study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2017-04-18 (Actual); Primary Completion 2017-06-23 (Actual); Study Completion 2017-06-23 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Concentration (Cmax) | Part 1: Pre-dose, 0.5 up to 48 hours post-dose Days 1, 9. Part 2: pre-dose, 0.5 up to 96 hours post-dose Days 1, 12. Part 3: pre-dose, 0.5 up to 48 hours post-dose on Days 1, 9. Part 4: pre-dose, 0.5 up to 48 hours post-dose Days 1, 10
  Cmax for midazolam (Part 1), rosuvastatin (Part 2), and simvastatin (Part 3) in the presence and absence of GDC-0853 and Cmax for GDC-0853 (Part 4) in the presence and absence of itraconazole.
Area Under the Concentration-Time Curve From Hour 0 to the Last Measurable Concentration (AUC0-t) | Part 1: Pre-dose, 0.5 up to 48 hours post-dose Days 1, 9. Part 2: pre-dose, 0.5 up to 96 hours post-dose Days 1, 12. Part 3: pre-dose, 0.5 up to 48 hours post-dose on Days 1, 9. Part 4: pre-dose, 0.5 up to 48 hours post-dose Days 1, 10
  AUC0-t for midazolam (Part 1), rosuvastatin (Part 2), and simvastatin (Part 3) in the presence and absence of GDC-0853 and AUC0-t for GDC-0853 (Part 4) in the presence and absence of itraconazole.

SECONDARY OUTCOMES:
Percentage of Participants with Adverse Events (AEs) and AEs of Special Interest (AESIs) | Up to approximately 7 weeks
  An AE is any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product, regardless of causal attribution. AESIs include any serious infection, any infections requiring intravenous antimicrobials, and any opportunistic infections; bleeding events of moderate or greater severity; a laboratory result of aspartate aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >5 × upper limit of normal (ULN) or an AST or ALT > 3 × ULN in combination with a total bilirubin > 2 × ULN, of which at least 35% is direct bilirubin or there is clinical jaundice; cases of potential drug-induced liver injury that include an elevated ALT or AST in combination with either an elevated bilirubin or clinical jaundice, as defined by Hy's law; or suspected transmission of an infectious agent by the study drug.
Cmax | 0.5 up to 12 hours post-dose on Days 11 and 12
  Cmax for GDC-0853 (Parts 2 and 3) in the presence and absence of rosuvastatin and simvastatin, respectively, and Cmax for itraconazole (Part 4) in the presence and absence of GDC-0853.
AUC0-12 | 0.5 up to 12 hours post-dose on Days 11 and 12
  AUC0-12 for GDC-0853 (Parts 2 and 3) in the presence and absence of rosuvastatin and simvastatin, respectively, and AUC0-12 for itraconazole (Part 4) in the presence and absence of GDC-0853.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (3):
- United States (3):
  - Covance Research Unit - Daytona, Daytona Beach, Florida
  - Covance Clinical Research Unit Inc.; Covance Gfi Research, Evansville, Indiana
  - Covance Clinical Research Unit, Inc, Madison, Wisconsin